CLINICAL TRIAL: NCT01812681
Title: Is Higher Cord Blood 25(Oh)-Vitamin D Level Preventive For Any Morbidity Including Rds, Pda, Nec, Bpd And Rop In Preterm Infants
Brief Title: Cord Blood 25(oh)-Vitamin D Level in Preterm Infants and Associated Morbidities
Status: Completed | Type: Observational
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Serdar Beken, MD, Dr. Sami Ulus Children's Hospital
Other Study IDs: B.10.4.İSM.4.06.68.49; B.10.4.İSM.4.06.68.49 (Other: Ethics Committe)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: vitamin D, Respiratory distress syndrome, sepsis, preterm
MeSH Terms: conditions — Respiratory Distress Syndrome; Sepsis; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low vitamin D level: The premature infants with low cord blood vitamin D level
- Normal Vitamin D: The premature infants with normal vitamin D level

SUMMARY:
Experimental and observational studies have shown that vitamin D deficiency may be associated with an increased risk for non-bone diseases and/or abnormal development for the other systems of fetus. The aim of this study is to determine the relationship between cord blood 25-hydroxyvitamin D (25 (OH) D) concentrations and the subsequent risk of morbidities including RDS, PDA, NEC, BPD AND ROP in preterm infants.

DETAILED DESCRIPTION:
It was shown that vitamin D play important role in the pathogenesis of long term morbidities of newborn. Experimental and observational studies have shown that vitamin D deficiency may be associated with an increased risk for non-bone diseases and/or abnormal development for the other systems of fetus. The aim of this study is to determine the relationship between cord blood 25-hydroxyvitamin D (25 (OH) D) concentrations and the subsequent risk of morbidities including RDS, PDA, NEC, BPD AND ROP in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* infants <32 weeks of gestational age

Exclusion Criteria:

* infants with major congenital abnormality
* infants >32 weeks of gestational age

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Dilli, Assoc Prof, Study Director — Sami Ulus CH
Locations (1):
- Sami Ulus CH, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Grant WB. Vitamin D supplementation of mother and infant could reduce risk of sepsis in premature infants. Early Hum Dev. 2010 Feb;86(2):133. doi: 10.1016/j.earlhumdev.2010.02.003. Epub 2010 Feb 25. No abstract available. PMID 20188500
- [Derived] Fettah ND, Zenciroglu A, Dilli D, Beken S, Okumus N. Is higher 25-hydroxyvitamin D level preventive for respiratory distress syndrome in preterm infants? Am J Perinatol. 2015 Feb;32(3):247-50. doi: 10.1055/s-0034-1383849. Epub 2014 Sep 13. PMID 25217734

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Vitamin D Level | Normal Vitamin D
Started | 60 | 24
Completed | 57 | 24
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Vitamin D Level | Normal Vitamin D | Total
Number analyzed (Participants) | 57 | 24 | 81
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 27.9 (2.4) | 29.2 (1.8) | 28.3 (3.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57 | 24 | 81
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 12 | 45
  Male | 24 | 12 | 36
Region of Enrollment [Number; unit: participants]
  Turkey | 57 | 24 | 81

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Distress Syndrome
Description: The association of vitamin D level with respiratory distress syndrome
Time Frame: three days
Measure: Number; unit: participants
Arm/Group | Low Vitamin D Level | Normal Vitamin D
Number analyzed (Participants) | 57 | 24
participants | 52 | 3

2. Secondary Outcome: Sepsis
Description: Association of vitamin D level with sepsis
Time Frame: four weeks
Measure: Number; unit: participants
Arm/Group | Low Vitamin D Level | Normal Vitamin D
Number analyzed (Participants) | 57 | 24
participants | 18 | 3

ADVERSE EVENTS:
Arm/Group | Low Vitamin D Level | Normal Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/24
Other Adverse Events (participants affected / at risk) | 0/57 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No